CLINICAL TRIAL: NCT04433689
Title: Change in Corneal Biomechanics During Pregnancy
Brief Title: Corneal Biomechanics During Pregnancy
Acronym: CorvisPreg
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: CorvisPreg
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Pregnancy
Keywords: pregnancy; corneal biomechanical properties; intraocular pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant woman, age 18 to 38 yo, with uncomplicated singleton pregnancy and no ocular diseases.
  Interventions: Device: Non-Contact measurement of corneal properties

INTERVENTIONS:
Device: Non-Contact measurement of corneal properties — Corneal Properties will be measurement with the non-contact Corvis ST Air-Puff Tonometer by Oculus Inc.

SUMMARY:
It is known that intraocular pressure changes during pregnancy. Collagen structure changes during pregnancy to enable softening of the symphysis, whitening of the birth chanel, and, thus, ultimately to enable delivery of a child. The cornea consists of highly structured collagen fibers. Hence, it seams logically that corneal biomechanics also change during pregnancy.

DETAILED DESCRIPTION:
It is known that intraocular pressure changes during pregnancy. Collagen structure changes during pregnancy to enable softening of the symphysis, whitening of the birth chanel, and, thus, ultimately to enable delivery of a child. The cornea consists of highly structured collagen fibers. Hence, it seams logically that corneal biomechanics also change during pregnancy.

Measurement of intraocular pressure is highly dependant on corneal properties. With the Corvis ST device by Ocular Inc. it is possible to measure intraocular pressure and investigated corneal biomechanics. The aim of this study is therefore to compare corneal biomechanical properties during the third trimester with corneal biomechanical properties at 3 months after delivery.

ELIGIBILITY:
Inclusion Criteria:

* females
* pregnant
* age 18 to 38 yo
* uncomplicated singleton pregnancy

Exclusion Criteria:

* any history of ocular disease or surgery other than conjunctivitis, especially no history of glaucoma or corneal disease
* systemic diseases, i.e. diabetes, hypertension, collagenase
* current contact lens wear
* before pregnancy taking any systemic or ocular medications

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Study Population: healthy pregnant women with uncomplicated singleton pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Deformation Amplitude | at 3 month post delivery compared to during third trimester
  Change in Deformation Amplitude (in millimeters) at 3 month post delivery compared to during third trimester will be assessed.
Change in Applanation Length | at 3 month post delivery compared to during third trimester of the pregnancy
  Change in Applanation Length (in millimeters) at 3 month post delivery compared to during third trimester of the pregnancy will be assessed.
Change in Corneal Velocity | at 3 month post delivery compared to during third trimester of the pregnancy
  Change in Corneal Velocity (in meters/second) at 3 month post delivery compared to during third trimester of the pregnancy will be assessed.
Change in corneal thickness | at 3 month post delivery compared to during third trimester of the pregnancy
  Change in corneal thickness (in millimeters) at 3 month post delivery compared to during third trimester of the pregnancy will be assessed.
Change in Intraocular pressure | at 3 month post delivery compared to during third trimester of the pregnancy
  Change in intraocular pressure (in millimeters of mercury, mmHg) at 3 month post delivery compared to during third trimester of the pregnancy will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Toeteberg-Harms, MD, FEBO, Principal Investigator — University Hospital Zurich, Dpt. of Ophthalmology
Locations (1):
- Department of Ophthalmology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No